CLINICAL TRIAL: NCT06461455
Title: Clinical Performance Evaluation of Two Frequent Replacement Silicone Hydrogel Multifocal Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLR624-C001
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Presbyopia; Astigmatism
Keywords: Myopia; Hyperopia; Multifocal; Toric
MeSH Terms: conditions — Presbyopia; Astigmatism; Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LID230451, then ULTRA MFfA (Other): Lehfilcon A multifocal for astigmatism contact lenses worn in Period 1, followed by samfilcon A multifocal for astigmatism contact lenses worn in Period 2, as randomized. The study lenses will be worn bilaterally (in both eyes) during typical contact lens wearing hours for at least 8 hours per day during each wear period [30 days (-2/+1)]. Study lenses will be removed daily for cleaning and disinfection with CLEAR CARE.
  Interventions: Device: Lehfilcon A multifocal for astigmatism contact lenses; Device: Samfilcon A multifocal for astigmatism contact lenses; Device: CLEAR CARE® Cleaning & Disinfecting Solution
- ULTRA MFfA, then LID230451 (Other): Samfilcon A multifocal for astigmatism contact lenses worn in Period 1, followed by lehfilcon A multifocal for astigmatism contact lenses worn in Period 2, as randomized. The study lenses will be worn bilaterally (in both eyes) during typical contact lens wearing hours for at least 8 hours per day during each wear period [30 days (-2/+1)]. Study lenses will be removed daily for cleaning and disinfection with CLEAR CARE.
  Interventions: Device: Samfilcon A multifocal for astigmatism contact lenses; Device: Lehfilcon A multifocal for astigmatism contact lenses; Device: CLEAR CARE® Cleaning & Disinfecting Solution

INTERVENTIONS:
Device: Lehfilcon A multifocal for astigmatism contact lenses — Investigational multifocal contact lenses for astigmatism
  Arms: LID230451, then ULTRA MFfA
Device: Samfilcon A multifocal for astigmatism contact lenses — Commercially available multifocal contact lenses for astigmatism
  Other Names: ULTRA® Multifocal for Astigmatism
Device: CLEAR CARE® Cleaning & Disinfecting Solution — Hydrogen peroxide-based contact lens cleaning and disinfection system
  Other Names: CLEAR CARE
  Arms: LID230451, then ULTRA MFfA
Device: Lehfilcon A multifocal for astigmatism contact lenses — Investigational multifocal contact lenses for astigmatism
  Arms: ULTRA MFfA, then LID230451
Device: CLEAR CARE® Cleaning & Disinfecting Solution — Hydrogen peroxide-based contact lens cleaning and disinfection system
  Other Names: CLEAR CARE
  Arms: ULTRA MFfA, then LID230451

SUMMARY:
The purpose of this study is to evaluate on-eye clinical performance of the investigational contact lenses following 30 days of wear in the intended population.

DETAILED DESCRIPTION:
Subjects will wear two different contact lens study products in a cross-over fashion. Each study product type will be worn for approximately 30 days. A washout period of 2-4 days will occur prior to the first wear period and between the two wear periods. Subjects will be expected to attend 5 office visits. The total duration of study participation is approximately 66 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Habitual wearer of biweekly/monthly replacement soft multifocal or multifocal toric contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months;
* Manifest cylinder equal to or greater than 0.75 diopter (D) in each eye at Screening;
* Willing to not use readers while wearing study contact lenses for duration of the study;
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Use of topical ocular medications and artificial tear or rewetting drops that would require instillation during contact lens wear;
* Wears habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment;
* Monovision contact lens wearers and wearers of contact lens in one eye only;
* Other protocol-defined exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (11):
- United States (11):
  - Dr.Elsa Pao, O.D, Oakland, California
  - Pacific Rims Optometry, San Francisco, California
  - Drs. Giedd, P.A., Maitland, Florida
  - Vision Health Institute, Orlando, Florida
  - Kannarr Eye Care LLC, Pittsburg, Kansas
  - Wesley Optometric Consulting, Medina, Minnesota
  - Oculus Research, Inc., Garner, North Carolina
  - ProCare Vision Centers, Inc., Granville, Ohio
  - Insight Research Clinic LLC, Powell, Ohio
  - Optometry Group, PLLC, Memphis, Tennessee
  - Dawn M. Rakich, OD, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 11 investigative sites.
Pre-assignment Details: Of the 95 enrolled, 6 subjects were discontinued as screen failures prior to randomization, and 4 subjects were discontinued post randomization and prior to exposure to the study lenses. This reporting group includes all subjects exposed to any study lenses evaluated in this study.
Groups:
- LID230451, Then ULTRA MFfA: Lehfilcon A multifocal for astigmatism contact lenses worn in Period 1, followed by samfilcon A multifocal for astigmatism contact lenses worn in Period 2, as randomized. The study lenses were worn bilaterally (in both eyes) during typical contact lens wearing hours for at least 8 hours per day during each wear period [30 days (-2/+1)]. Study lenses were removed daily for cleaning and disinfection with CLEAR CARE.
- ULTRA MFfA, Then LID230451: Samfilcon A multifocal for astigmatism contact lenses worn in Period 1, followed by lehfilcon A multifocal for astigmatism contact lenses worn in Period 2, as randomized. The study lenses were worn bilaterally (in both eyes) during typical contact lens wearing hours for at least 8 hours per day during each wear period [30 days (-2/+1)]. Study lenses were removed daily for cleaning and disinfection with CLEAR CARE.
Period: First Wear Period (Approx 30 Days)
Arm/Group | LID230451, Then ULTRA MFfA | ULTRA MFfA, Then LID230451
Started | 46 | 39
Completed | 45 | 38
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Screen failure | 1 | 0
Period: Washout Period (Approx 2-4 Days)
Arm/Group | LID230451, Then ULTRA MFfA | ULTRA MFfA, Then LID230451
Started | 45 | 38
Completed | 45 | 37
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Second Wear Period (Approx 30 Days)
Arm/Group | LID230451, Then ULTRA MFfA | ULTRA MFfA, Then LID230451
Started | 45 | 37
Completed | 45 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects exposed to any study lenses evaluated in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | LID230451, Then ULTRA MFfA | ULTRA MFfA, Then LID230451 | Total
Number analyzed (Participants) | 46 | 39 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (9.4) | 55.9 (9.4) | 55.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 56
  Male | 17 | 12 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 39 | 27 | 66
  Black or African American | 2 | 2 | 4
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 10 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 46 | 39 | 85

OUTCOME MEASURES:

1. Primary Outcome: Mean Binocular Visual Acuity at Distance (4 Meters) at Day 30 With Study Lenses
Description: Visual Acuity (VA) was assessed at a distance of 4 meters with both eyes together (binocular) under high contrast, high illumination lighting with study lenses in place. VA was measured using letter charts and recorded in the logarithm of the minimum angle of resolution (LogMAR). A LogMAR value of 0 equates to 20/20 Snellen VA (normal distance eyesight), with negative LogMAR values representing better than 20/20 VA. The LogMAR VA scale ranges from -0.30 (20/10 Snellen) to 1.00 (20/200 Snellen).
Time Frame: Day 30 (-2/+1) of each wear period. A wear period was 30 days (-2/+1) according to randomization assignment.
Population: Full Analysis Set with data at visit
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- LID230451: Lehfilcon A multifocal for astigmatism contact lenses worn in Period 1 or Period 2, as randomized. The study lenses were worn bilaterally (in both eyes) during typical contact lens wearing hours for at least 8 hours per day during each wear period [30 days (-2/+1)]. Study lenses were removed daily for cleaning and disinfection with CLEAR CARE.
- ULTRA MFfA: Samfilcon A multifocal for astigmatism contact lenses worn in Period 1 or Period 2, as randomized. The study lenses were worn bilaterally (in both eyes) during typical contact lens wearing hours for at least 8 hours per day during each wear period [30 days (-2/+1)]. Study lenses were removed daily for cleaning and disinfection with CLEAR CARE.
Arm/Group | LID230451 | ULTRA MFfA
Number analyzed (Participants) | 82 | 81
logMAR | -0.50 (0.10) | -0.08 (0.09)
Statistical Analysis 1: Comparison: LID230451 vs ULTRA MFfA; Test type: Non-Inferiority — Non-inferiority in distance VA was declared if upper confidence limit was less than 0.05; Since a non-inferiority hypothesis is being tested, confidence limit is more appropriate than p-value in assessing the results against the predefined non-inferiority margin; Least Squares Mean Difference = -0.05, 95% CI 1-sided [upper limit 0.04], Standard Error of Mean 0.011 — LSM results based on mixed effects repeated measures model with both fixed (lens, visit, lens by visit interaction, period, and lens sequence) and random (subject) effects. Difference=LID230451-ULTRA MFfA. Sign is retained with the rounded value

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from time of consent to study exit, approximately 66 days. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects exposed to any study lenses evaluated in this study, as treated.
Description: All subjects were monitored for serious and other ocular and nonocular AEs. However, the nonocular AE arms were not considered at Risk for ocular adverse event terms as the arms are reporting nonocular-specific AEs. Similarly, the ocular AE arms were not considered at Risk for nonocular adverse event terms as the arms are reporting ocular-specific AEs. All-Cause Mortality was not monitored for the ocular arms.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study lenses.
- LID230451 Ocular; LID230451 Nonocular: Events reported in this group occurred while exposed to the lehfilcon A multifocal for astigmatism contact lenses.
- ULTRA MFfA Ocular; ULTRA MFfA Nonocular: Events reported in this group occurred while exposed to the samfilcon A multifocal for astigmatism contact lenses.
Arm/Group | Pretreatment | LID230451 Ocular | LID230451 Nonocular | ULTRA MFfA Ocular | ULTRA MFfA Nonocular
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/0 | 0/83 | 0/0 | 0/84
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/166 | 0/83 | 0/168 | 0/84
Other Adverse Events (participants affected / at risk) | 0/85 | 0/166 | 0/83 | 0/168 | 0/84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT06461455/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT06461455/SAP_001.pdf